CLINICAL TRIAL: NCT00371878
Title: Open Label Study of Lung and Serum Immunoglobulin Responses to 7-Valent Pneumococcal Conjugate Vaccine in HIV Infected and Non-HIV Infected Malawian Adults
Brief Title: Immunogenicity of 7-Valent Pneumococcal Conjugate Vaccine in Lung Fluid of Adults With and Without HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Liverpool University Hospital (Other Government)
Collaborators: Kamuzu University of Health Sciences (Other); Liverpool School of Tropical Medicine (Other); Wellcome Trust (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BAL0601; ISRCTN54494731; ISRCTN 061230; P99/00/101; P99/00/102
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2006-09

CONDITIONS: Pneumonia; Meningitis; Invasive Pneumococcal Disease; HIV
Keywords: Vaccine; Lung; Bronchoalveolar lavage; Lymphocyte; Immunoglobulin; HIV; Streptococcus pneumoniae; Conjugate vaccine
MeSH Terms: conditions — Pneumonia; Meningitis | interventions — Heptavalent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 7-valent pneumococcal conjugate vaccine (Prevnar)

SUMMARY:
Lung immune responses are regulated independently of systemic responses. Injected vaccines may induce optimal responses in blood but not at mucosal surfaces. We compared the responses in serum and lung fluid to injected pneumococcal conjugate vaccine.

DETAILED DESCRIPTION:
We tested the hypothesis that conjugate vaccine offered less protection against pneumonia due to a reduced mucosal response compared to serum. We further hypothesized that this response would be further compromised with HIV co-infection[32] due to lack of local CD4 lymphocyte support and an altered alveolar milieu. We measured pneumococcal capsular specific immunoglobulin responses to 7-valent conjugate vaccine in both lung fluid and serum from healthy HIV infected and uninfected volunteers, together with flow cytometric assessment of the relative numbers and phenotypes of BAL T lymphocyte, B lymphocyte and macrophages.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer adults

Exclusion Criteria:

* pregnant, recent illness, previous vaccination, asthma

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-02; Study Completion 2003-10

PRIMARY OUTCOMES:
Immunoglobulin titres in bronchoalveolar fluid

SECONDARY OUTCOMES:
Immunoglobulin titres in serum
Lung lymphocyte phenotype
HIV viral load

CONTACTS AND LOCATIONS:
Overall Officials: Neil French, PhD FRCP, Study Director — Karonga Prevention Study, London School of Tropical Medicine and Hygience; Stephen B Gordon, MA MD FRCP, Principal Investigator — Liverpool School of Tropical Medicine, Liverpool, UK
Locations (1):
- Wellcome Trust Laboratories and Dept of Medicine, Queen Elizabeth Central Hospital, Blantyre, Malawi